CLINICAL TRIAL: NCT02050659
Title: Omentectomy in Radical Gastrectomy for Gastric Cancer Trial
Acronym: OMEGA
Status: Completed | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Responsible Party: Principal Investigator, S.S. Gisbertz, MD PhD, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: OMEGA
Record Dates: First submitted 2014-01-28; First posted 2014-01-31 (Estimated); Last update posted 2015-03-10 (Estimated); Status verified 2015-03

CONDITIONS: Omentum; Stomach Neoplasms
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
In patients with gastric cancer, traditionally a complete omentectomy is performed as part of a radical gastrectomy with a modified D2 lymph node dissection. The omentectomy increases operation time significantly, especially in laparoscopic procedures. Patients remain more vulnerable for peritoneal infections and intestinal adhesions following omentectomy. Furthermore one can debate whether a complete omentectomy is indicated from an oncologic viewpoint. In the present study we prospectively evaluated the presence of tumor load in the greater omentum of patients with potentially curative gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* an in potentially curative gastric cancer
* age > 18 year

Exclusion Criteria:

* palliative resection
* age < 18 year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with a castric carcinoma who received an in potentially curative gastric resection
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2012-03; Primary Completion 2014-01 (Actual); Study Completion 2014-02 (Actual)

PRIMARY OUTCOMES:
tumorload in the greater omentum | at the time of pathologic investigation

CONTACTS AND LOCATIONS:
Locations (1):
- Academic Medical Centre, Amsterdam, Netherlands

REFERENCES:
- [Derived] Jongerius EJ, Boerma D, Seldenrijk KA, Meijer SL, Scheepers JJ, Smedts F, Lagarde SM, Balague Ponz O, van Berge Henegouwen MI, van Sandick JW, Gisbertz SS. Role of omentectomy as part of radical surgery for gastric cancer. Br J Surg. 2016 Oct;103(11):1497-503. doi: 10.1002/bjs.10149. Epub 2016 Aug 23. PMID 27550526